CLINICAL TRIAL: NCT02982317
Title: Automated UltraSound Software for Identification of Lumbar Vertebral Levels in Obstetric Patients
Brief Title: Automated UltraSound Software for Identification of Lumbar Vertebral Levels
Acronym: AUSSI
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anton Chau, PI, University of British Columbia
Other Study IDs: H16-02858
Record Dates: First submitted 2016-11-15; First posted 2016-12-05 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Anesthesia
Keywords: Neuraxial anesthesia; Obstetrics; Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: All patients recruited will undergo the same protocol. An anesthesiologist will perform manual palpation of the patients lumbar spine and identification of the intervertebral spaces from L1-S1. A member of the UBC Department of Engineering will perform the US scanning and level identification using the novel US technology. In addition, freehand US will be used by two practitioners to determine the participant's lumbar level locations as per gold standard.
  Interventions: Procedure: Manual palpation identification lumbar spine; Procedure: Automated ultrasound technology identification; Procedure: Lumbar level identification gold standard ultrasound

INTERVENTIONS:
Procedure: Manual palpation identification lumbar spine
Procedure: Automated ultrasound technology identification — This technology involves a standard ultrasound machine and curvilinear probe- what is novel is the software which will be connected to the ultrasound machine
Procedure: Lumbar level identification gold standard ultrasound

SUMMARY:
A novel automated ultrasound software system has been developed which identifies for the practitioner the intervertebral spaces in the lumbar area. This study aims to investigate whether this new technology has a greater accuracy of identifying intervertebral spaces that manual palpation.

DETAILED DESCRIPTION:
The use of ultrasound is one of the most accurate ways to identify the correct vertebral level for needle insertion in spinal/epidural anesthetics, however this is not commonly used. A novel automated ultrasound software system has been developed by the UBC Department of Engineering which identifies for the practitioner the intervertebral spaces in the lumbar area. This study aim to investigate whether this new technology has a greater accuracy of identifying intervertebral spaces that manual palpation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* ≥ 19 years old
* Term pregnancy (≥ 37 weeks gestation age)
* Scheduled for elective Cesarean section
* Ability to read English in order to understand the consent form

Exclusion Criteria:

* Patient refusal to participate
* BMI ≥ 40
* Scoliosis
* Previous lower back surgery or known spinal abnormalities
* Inability to palpate bony landmarks in lumbar region
* Active labour (cervical dilatation >5cm)
* Allergy to epidural tape, surgical paper tape, or felt pen

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Parturients scheduled for an elective Cesarean section at BC Women's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of identifying L3/L4 of agreement between the two techniques against the freehand US (control) | Within 1 hour of recuitment

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD, Principal Investigator — Univeristy of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hetherington J, Brohan J, Rohling R, Gunka V, Abolmaesumi P, Albert A, Chau A. A novel ultrasound software system for lumbar level identification in obstetric patients. Can J Anaesth. 2022 Oct;69(10):1211-1219. doi: 10.1007/s12630-022-02300-6. Epub 2022 Aug 9. PMID 35941333